CLINICAL TRIAL: NCT05281796
Title: Gingival Crevicular Fluid And Salivary Levels of Galectin-3 in Patients With Gingivitis And Patients With Stage III Periodontitis: An Observational Study
Brief Title: Evaluation of Galectin-3 Levels in GCF And Saliva of Patients With Different Periodontal Diseases
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed saad arafa ali, Principal Investigator mohamed saad, Cairo University
Other Study IDs: 1512022
Record Dates: First submitted 2022-03-07; First posted 2022-03-16 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Periodontal Diseases
Keywords: galectin-3
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- healthy patient: Full-mouth clinical periodontal measurements recorded, saliva and GCF obtained
  Interventions: Diagnostic Test: GCF obtaining; Diagnostic Test: saliva obtaining
- gingivitis patient: Full-mouth clinical periodontal measurements recorded, saliva and GCF obtained
  Interventions: Diagnostic Test: GCF obtaining; Diagnostic Test: saliva obtaining
- patients with Stage III periodontitis: Full-mouth clinical periodontal measurements recorded, saliva and GCF obtained
  Interventions: Diagnostic Test: GCF obtaining; Diagnostic Test: saliva obtaining

INTERVENTIONS:
Diagnostic Test: GCF obtaining — GCF sample collection by Enzyme-Linked Immunosorbent Assay (ELISA)
Diagnostic Test: saliva obtaining — Saliva sample collection by Enzyme-Linked Immunosorbent Assay (ELISA)

SUMMARY:
The aim of this study is to assess the levels of galectin-3 in the GCF and saliva in patient with gingivitis and patient with stage III periodontitis.

DETAILED DESCRIPTION:
The aim of this study is to assess the levels of galectin-3 in the GCF and saliva in patient with gingivitis and patient with stage III periodontitis.

This study will be conducted in the Oral Medicine and Periodontology department, Faculty of Dentistry- Cairo University, Egypt.

Patients will be selected from the outpatient clinic of the department of Oral Medicine and Periodontology, Faculty of Dentistry-Cairo University.

ELIGIBILITY:
Inclusion Criteria:

1. For healthy group: individuals with less than 10% bleeding on probing area, having a probing depth less than 4mm and no loss of attachment were included in the study.
2. For the gingivitis group: individuals with 10% or more bleeding on probing area, having a probing depth of less than 4mm and no attachment loss.
3. For the periodontitis group that has not received periodontal treatment in the last 6 months
4. For the periodontitis group: individuals with 30% or more bleeding on probing area, at least 2 teeth not adjacent to each quarter jaw with a depth of 5 mm or more and 4 mm or more attachment loss, coronal 1/3 and more on radiography (horizontal and / or vertical) bone loss.
5. Presence of a minimum of 15 natural teeth.

Exclusion Criteria:

1. Individuals with any known systemic disease.
2. Pregnant and lactating women.
3. Individuals that received periodontal treatment within the last 6 months.
4. Individuals with a history of systemic antibiotics and anti-inflammatory drugs within the last 3 months.
5. Former or current smokers.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Dental patients will be recruited in a consecutive manner from the clinic of the department of Oral Medicine and Periodontology, Faculty of Dentistry - Cairo University. Medical history and dental history will be taken; thorough oral examination will be done. The aim of the study will be explained to the patient and the patient's acceptance to participate in the survey will be received. Nonrespondent patients or patients refusing to participate will be reported with the cause of their refusal. Conventional oral and periodontal examination will be held on a dental unit using the light of the unit, mirror and probe
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2022-01-22 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
galectin-3 in GCF | 24 hours after taking the clinical measurements at the first visit
  The total amount of Galectin-3 in GCF
galectin-3 in saliva. | 24 hours after taking the clinical measurements at the first visit
  The total amount of Galectin-3 in saliva

SECONDARY OUTCOMES:
Pocket depth | 24 hours before taking GCF and salivary samples
  in mm
Clinical attachment level | 24 hours before taking GCF and salivary samples
  in mm
Bleeding on Probing | 24 hours before taking GCF and salivary samples
  By gently probing the orifice of the gingival crevice, the periodontal probe will be inserted 1 to2 mm into the gingival sulcus starting at one interproximal area and moving to the other. If bleeding occurs within 10 seconds a positive finding is recorded.
Plaque Index | 24 hours before taking GCF and salivary samples
  Scores: 0: No plaque
  1. A film of plaque adhering to the free gingival margin and adjacent area of the tooth. The plaque may be seen insitu only after application of a disclosing solution or by using the probe on the tooth surface.
  2. Moderate accumulation of soft deposit s within the gingival pocket, or the tooth and gingival margin, which can be seen with the naked eye.
  3. Abundance of soft matter within the gingival pocket and/or on the tooth and gingival margin.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Sa Ali, master's, Principal Investigator — Cairo University
Locations (1):
- Cairo university Faculty of dentistry, Cairo, Egypt